CLINICAL TRIAL: NCT06312046
Title: Motor-cognitive Performance in People With Multiple Sclerosis - Brain Activity and Effects of Balance Exercise
Brief Title: Motor-cognitive Performance in People With Multiple Sclerosis
Acronym: HiBalance-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Sverker Johansson, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018 374-31
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Postural Balance
Keywords: Balance; Exercise; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcome assessor will not participate in the provided training program. Care provider will not perform the analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Balance training intervention group (Experimental): The program HiBalance-MS is based on scientifically well-established principles of exercise training and postural control. It will be conducted as a progressive individually adjusted group training to challenge the specific balance deficit of every participant. To ensure highly challenging exercises, each task is individually adjusted, e.g., by altering the base of support, increasing speed, restricting vision and varying grade of multitasking. Daily variation in capacity will be rated before each training session and participants will at the end of each session rate the challenging level. The training will be performed in the clinic, at Karolinska University Hospital, for an hour, twice a week for 10 weeks, as a group intervention including 6 to 8 participants and facilitated by two physiotherapists/trainers.
  Interventions: Other: HiBalance-MS
- No intervention control group (No Intervention): Participants in the control group are encouraged to maintain their normal physical activities and are not restricted from participation in ongoing rehabilitation programs.

INTERVENTIONS:
Other: HiBalance-MS — See arm description for intervention group.
  Arms: Balance training intervention group

SUMMARY:
Having a neurological disease such as multiple sclerosis (MS) leads to difficulties in balance and gait with or without concurrent performance of cognitive tasks, hindering activity performance and influencing the possibilities for an independent lifestyle.

The investigators have adapted a previously developed balance training program to a highly challenging program specifically directed to MS (HiBalance-MS). This program was recently tested and found feasible in a pilot study. The investigators will now perform a randomized controlled trial in people with MS, in order to determine the effects of the program. The hypothesis is that progressively challenging balance exercise programs that are specific to the balance control domains affected by MS will be effective to improve balance control, walking, motor-cognitive performance, activity performance and health related quality of life.

DETAILED DESCRIPTION:
Everyday living means being in complex environments and performing complex activities which usually consist of and require a combination of motor and cognitive skills. Having a neurological disease such as multiple sclerosis (MS) compromises the motor-cognitive performance. This leads to difficulties in balance and gait with or without concurrent performance of cognitive tasks, hindering activity performance and influencing the possibilities for an independent lifestyle.

The investigators have, in a co-design process with stakeholders, adapted a HiBalance program, originally developed by the Franzén research group for people with Parkinson's disease and combining motor-cognitive exercises in a progressively more difficult manner (HiBalance-PD), to a program specifically developed to MS (HiBalance-MS). The developed HiBalance-MS program was recently tested and found feasible in a pilot study (results published 2023). The investigators will now perform a randomized controlled trial in people with MS, in order to determine the effects of a highly challenging balance training program (HiBalance-MS) on physical and cognitive functioning, and activity performance, in this group. The results will have immediate application and clinical relevance. With improved balance control people with MS will also gain other health benefits related to an active lifestyle and a better everyday life.

The hypothesis that motor-cognitive performance is reduced and impact activity performance in people with MS. They also hypothesize that progressively challenging balance exercise programs that are specific to the balance control domains affected by MS will be effective to improve balance control, walking, motor-cognitive performance, activity performance and health related quality of life.

Participants will be recruited through Karolinska University Hospital, through physiotherapists and physicians specialized in neurology in Stockholm and via advertisement in newspapers and the patient organization NEURO Sweden. According to earlier power calculations for detecting effects in balance and gait measures after this particular intervention, the investigators anticipate 40 to 50 participants in each group to detect significant changes.

The HiBalance-MS program is based on scientifically well-established principles of exercise training and postural control. It will be conducted as a progressive individually adjusted group training to challenge the specific balance deficit of every participant. Four main sub-systems underlying balance control (stability limits, anticipatory postural adjustments, sensory integration and motor agility) are used to target specific balance impairments. To ensure highly challenging exercises, each task is individually adjusted. Daily variation in capacity will be rated before each training session and participants will at the end of each session rate the challenging level. The training will be performed in the clinic (Karolinska University hospital) for an hour, twice a week for 10 weeks, as a group intervention (6 to 8 participants) facilitated by two physiotherapists/trainers.

ELIGIBILITY:
Inclusion Criteria:

* an MS diagnosis according to McDonald criteria;
* an overall MS-disability score from 2.0 to 5.5 according to the Expanded Disability Status Scale;
* ability to walk 100 m without aid;
* a maximum score of 24 in the Mini-BESTest (i.e., < 25 points)
* 18 to 65 years of age

Exclusion Criteria:

* cognitive impairment as indicated by a score <21 in the Montreal Cognitive Assessment;
* presence of other conditions that would substantially influence balance;
* an MS relapse or change of disease-modifying treatment within the past 8 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Mini Balance Evaluation Systems test. | Pre intervention baseline and post intervention at 10 weeks.
  Balance performance. A rating scale for dynamic balance incorporating 14 different balance and gait items that are assessed by a physical therapist on a scale from 0-2. Points between 0 and 28; a higher total score indicates better balance control.

SECONDARY OUTCOMES:
10-Meter Walk Test, maximum speed. | Pre intervention baseline and post intervention at 10 weeks.
  Gait performance. Maximum gait speed (meter/second), a higher score indicates higher gait speed.
10-Meter Walk Test, self-selected speed. | Pre intervention baseline and post intervention at 10 weeks.
  Gait performance. Self-selected comfortable gait speed (meter/second), a higher score indicates higher self-selected comfortable gait speed.
2-Minute Walk Test, self-selected speed. | Pre intervention baseline and post intervention at 10 weeks.
  Gait performance. Self-selected gait speed (meter/second), a higher score indicates higher self-selected endurance gait speed.
Gait speed during simultaneous dual task performance. | Pre intervention baseline and post intervention at 10 weeks.
  Gait speed (meter/second), will be analyzed during dual task walking with the Ambulatory Parkinson´s Disease Monitoring (APDM) mobility Lab system. Dual tasking during walking will be performed with the Auditory stroop task, a test of cognitive function, see below. A higher score indicates higher gait speed during dual tasking,
Stride length during dual task gait performance. | Pre intervention baseline and post intervention at 10 weeks.
  Stride length (meter) during gait will be analyzed during dual task walking with the Ambulatory Parkinson´s Disease Monitoring (APDM) mobility Lab system. Dual tasking during walking will be performed with the Auditory stroop task, a test of cognitive function, see below.Longer stride length indicates better control during walking,
Step time during dual task gait performance. | Pre intervention baseline and post intervention at 10 weeks.
  Step time during gait (seconds) will be analyzed during dual task walking with the Ambulatory Parkinson´s Disease Monitoring (APDM) mobility Lab system. Dual tasking during walking will be performed with the Auditory stroop task, a test of cognitive function, see below. Shorter step time indicates better control during walking,
Response errors in dual task cognitive performance | Pre intervention baseline and post intervention at 10 weeks.
  Dual task cognitive performance during walking will be performed with the Auditory stroop task, a test of cognitive flexibility in selective executive functions. Cognitive performance of the dual task will be assessed as errors in the response (numbers) to the Auditory stroop task. Data colllection is performed through wireless headphones (RazerTM ManO'War) using Audacity software (version 3.0.2).
Reaction time in dual task cognitive performance | Pre intervention baseline and post intervention at 10 weeks.
  Dual task cognitive performance during walking will be performed with the Auditory stroop task, a test of cognitive flexibility in selective executive functions. Cognitive performance of the dual task will be assessed as reaction time (seconds) in the Auditory stroop task. Data colllection is performed through wireless headphones (RazerTM ManO'War) using Audacity software (version 3.0.2).
Six-Spot Step Test. | Pre intervention baseline and post intervention at 10 weeks.
  A test of complex walking. The Six-Spot Step Test is a 5 meter test-field criss-cross walk pattern where the subject while walking is simultaneously kicking wooden blocks from marked circles in the field. Mean time (seconds) of four trials is calculated, shorter time indicates better complex walking performance.
Completion time in the Trail Making Test. | Pre intervention baseline and post intervention at 10 weeks.
  The Trail Making Test (from Delis-Kaplan Executive Function System) assesses attention and psychomotor processing speed. The time (seconds) to complete the test, connecting numbers and letters correctly, is registered. Shorter completion time indicates better attention and higher psychomotor processing speed.
Number of errors in the Trail Making Test. | Pre intervention baseline and post intervention at 10 weeks.
  The Trail Making Test (from Delis-Kaplan Executive Function System) assesses attention and psychomotor processing speed. The number of mistakes/errors is registered. Less number of mistakes/errors indicates better attention and higher psychomotor processing speed.
Immediate and delayed recall in the Ray Auditory Verbal Learning Test. | Pre intervention baseline and post intervention at 10 weeks.
  The Ray Auditory Verbal Learning Test assesses episodic memory. In this test 15 words is repeatedly (five times) read for the subject. The subject is asked to recall as many as possible. The subject is asked again after 30 minutes to recall as many words as possible. The test assesses immediate recall (number) and delayed recall (number) of words where higher number of immediate and delayed recalled words indicates better episodic memory.
Cognitive processing speed in the Symbol Digit Modalities Test. | Pre intervention baseline and post intervention at 10 weeks.
  The Symbol Digit Modalities Test assesses cognitive processing speed. The subject is asked to pair specific numbers with given symbols. The number of correctly paired numbers and symbols within 90 seconds is registered where a higher number indicates higher cognitive processing speed.
Cognitive function - composite measure of three cognitive tests. | Pre intervention baseline and post intervention at 10 weeks.
  Cognitive function will also be assessed as a composite measure of a cognitive test battery consisting of: Trail making Test (from Delis-Kaplan Executive Function System), testing attention and and psychomotor processing speed); Ray Auditory Verbal Learning Test, assessment of episodic memory; and Symbol Digit Modalities Test, assessment of cognitive processing speed. First, the scores of each of the three tests will be standardised into z-scores using pre-scores. Models using different test are compared. The model including all three tests and using the robust diagonally weighted least square estimation will be chosen based on fit values. Last, the z-scores of each test and person are multiplied with the factor loadings and added together to create a sum score for each person and time point. A higher value = greater executive functions.
Physical activity level. | Pre-and-post-intervention over four to seven days when awake.
  Assessment with accelerometer Actigraph GT3X+. Participants wear the accelerometer around the hip, attached slightly above the iliac crest with an elastic band. They wear the accelerometer in their daily life for seven consecutive days (minimum four days), only removing it when showering, bathing, swimming, and at night. As a proxy for the level of daily physical activity, the number of steps per day will be used, where a higher number indicates higher level of physical activity.
Physical activity level, self-reported. | Pre intervention baseline and post intervention at 10 weeks.
  Frändin & Grimby Scale, a self-reported questionnaire (score 1-6, higher score = higher physical activity level measured in hours,
Physical exercise habits, self-reported. | Pre intervention baseline and post intervention at 10 weeks.
  A question regarding physical exercise habits is included (from The Swedish Research Council). Score 1-6, A higher score indicates larger interval of minutes per week used for physical exercise.
The generic Walk-12 questionnaire. | Pre intervention baseline and post intervention at 10 weeks.
  Self assessment of walking ability with the generic Walk-12 questionnaire. A total of 12 questions, possibility to score from 1 to 5. Total score between12 and 60. A higher score indicates perceived more limited walking ability.
Falls Efficacy Scale - International. | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported questionnaire regarding falls efficacy, A total of 16 questions, score 1-4. Total score from 16 to 64 points, a higher total score = more concerned of falling.
Assesment of anxiety with the Hospital Anxiety and Depression Scale. | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported questionnaire assessing anxiety and depression. Total score from 0 to 28 points, 14 points each on the depression and anxiety parts respectively. Lower scores on the anxiety part indicates less anxiety.
Assesment of depression with the Hospital Anxiety and Depression Scale. | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported questionnaire assessing anxiety and depression. Total score from 0 to 28 points, 14 points each on the depression and anxiety parts respectively. Lower scores on the depression part indicates less depression.
Modified Fatigue Impact Scale. | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported questionnaire which measures impact of fatigue on physical, cognitive and psychosocial functioning, The scale consists of 21 items, scored from 0 to 4. Total score ranges from 0 to 84 points. Higher scores indicate larger impact of fatigue (total impact or impact in physical, cognitive and psychosocial functioning.
Occupational Gap Questionnaire. | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported questionnaire measuring participation in everyday activities. The questionnaire includes 30 questions regarding if an activity is performed and regarding if the person wants to perform the activity. Number of activities performed (higher scores = better) and number of wanted but not performed activities (higher scores = worse) are counted .
Acceptance of Chronic Health Condition scale. | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported questionnaire (10 questions scored on a 5 category Likert rating scale measuring acceptance of chronic health condition. Scores from 1 to 50), a higher score = higher level of acceptance.
Multiple Sclerosis Impact Scale - physical impact. | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported diagnose-specific questionnaire assessing health-related quality of life. A total of 29 items (20 physical and 9 psychological). Items are rated from 1 to 5. Total score ranges from 20 to 100 in physical impact. Higher total score = worse physical impact.
Multiple Sclerosis Impact Scale - psychological impact. | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported diagnose-specific questionnaire assessing health-related quality of life. A total of 29 items (20 physical and 9 psychological). Items are rated from 1 to 5. Total scores range from 9 to 45 in psychological impact. Higher total score = worse psychological impact.
Euroqol-5 Dimensions-5 Level (EuroQoL-5D-5L). | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported generic questionnaire measuring health-related quality of life. The questionnaire assesses five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels - higher level score = increased disability.
Euroqol Visual Analogue Scale (EQ VAS). | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported generic questionnaire measuring health-related quality of life. In addition to the five dimensions of health (as described above) the EuroQoL-5D-5L includes a vertical visual analogue scale (the EQ VAS), which records the patient's self-rated health on the vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' (100) and 'Worst imaginable health state' (0).
World Health Organization Disability Assessment Schedule, version 2.0. (WHODAS 2.0) | Pre intervention baseline and post intervention at 10 weeks.
  A self-reported questionnaire consisting of 12 questions assessing disability. Total score from12 to 60, a higher score = worse disability.

CONTACTS AND LOCATIONS:
Overall Officials: Sverker Johansson, Ph.D, Principal Investigator — Karolinska Institutet, org.nr 202100-2973
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are not publicly available due to Swedish and European Union personal data legislation but are available from the principal investigator on reasonable request. Any sharing of data will be regulated via a data transfer and user agreement with the recipient.
Time Frame: The investigators plan to share this when applicable on the Open Science Platform or similar.
Access Criteria: The datasets generated during and/or analysed during the current study are not publicly available due to Swedish and European Union personal data legislation but are available from the principal investigator on reasonable request. Any sharing of data will be regulated via a data transfer and user agreement with the recipient.

REFERENCES:
- See also: Publication: A highly challenging balance training intervention for people with multiple sclerosis: a feasibility trial — https://pubmed-ncbi-nlm-nih-gov.proxy.kib.ki.se/36922859/